CLINICAL TRIAL: NCT04884360
Title: A Randomised, Double-blind, Placebo-controlled, Phase III Study of Olaparib Maintenance Monotherapy in Participants With BRCA Wild Type Advanced High Grade Serous or Endometrioid Ovarian Cancer Following Response to Standard First-line Platinum-based Chemotherapy (MONO-OLA1)
Brief Title: D9319C00001- 1L OC Mono Global RCT
Acronym: MONO-OLA1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9319C00001; 2020-005960-68 (EudraCT Number)
Record Dates: First submitted 2021-04-20; First posted 2021-05-13 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer
Keywords: BRCA Wild Type;; Double-blind;; Randomized;; Placebo-controlled;
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Olaparib tablets 300 mg oral twice daily (n=238). (Experimental): Participants in Group A will receive olaparib tablets taken orally at a dose of 300 mg twice daily for up to 2 years or until objective radiological disease progression as per RECIST 1.1 as assessed by the investigator, whichever is earlier, and as long as in the investigator's opinion they are benefiting from treatment and do not meet any other discontinuation criteria.
  Interventions: Drug: Olaparib
- Group B: Placebo tablets 300 mg oral twice daily (n=118) (Placebo Comparator): Participants in Group B will receive matching placebo tablets taken orally at a dose of 300 mg twice daily for up to 2 years or until objective radiological disease progression as per RECIST 1.1 as assessed by the investigator, whichever is earlier, and as long as in the investigator's opinion they are benefiting from treatment and do not meet any other discontinuation criteria.
  Interventions: Other: Matching placebo

INTERVENTIONS:
Drug: Olaparib — Olaparib tablets 300 mg oral twice daily
  Arms: Group A: Olaparib tablets 300 mg oral twice daily (n=238).
Other: Matching placebo — Matching placebo tablets taken orally at a dose of 300 mg twice daily
  Arms: Group B: Placebo tablets 300 mg oral twice daily (n=118)

SUMMARY:
This is a Phase III, randomised, double-blind, placebo-controlled, multicentre, international study assessing the efficacy and safety of maintenance olaparib compared with placebo in BRCAwt participants with Stage III to IV high grade serous or endometroid ovarian cancer (including fallopian tube cancer or primary peritoneal cancer) who are in complete or partial response following treatment with standard first-line platinum-based chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants must be ≥18 years at the time of (pre-)screening
2. Histological and staging criteria:Female participants who must have histologically newly diagnosed high-grade serous or high-grade endometrioid ovarian cancer, fallopian tube cancer, or primary peritoneal cancer that is Stage III or IV according to the International FIGO 2014.
3. Participants are eligible if they fulfil any of the following surgical criteria:

   * Stage III: primary debulking surgery with macroscopic residual disease post-surgery, neoadjuvant chemotherapy, or inoperable.
   * Stage IV: primary debulking surgery regardless of residual disease, neoadjuvant chemotherapy, or inoperable.
4. Chemotherapy criteria:

   * Participants must have received platinum-based chemotherapy consisting of a minimum of 6 treatment cycles and a maximum of 9, however, if platinum-based therapy must be discontinued early as a result of toxicities specifically related to the platinum regimen, participants must have received a minimum of 4 cycles of the platinum regimen.
   * Participants must have, in the opinion of the investigator, clinical CR or PR as per RECIST 1.1 criteria with no measurable lesion > 2 cm on the post-treatment scan and have no clinical evidence of disease progression or a rising CA-125 level (see inclusion criterion 5), following completion of this chemotherapy course.
   * A participant who received interval debulking surgery must have had ≥ 2 postoperative cycles of platinum-based therapy.
5. Participants must meet one of the criteria specified below for pre-treatment CA-125 measurements as follows:

   * CA-125 in the normal range or
   * CA-125 decrease by ≥ 90% during their front-line therapy that is stable for at least 7 days (ie, no increase > 15% from nadir). During screening, if the first CA-125 value is greater than the upper limit of normal (ULN), a second assessment must be performed at least 7 days after the first. If the second assessment is > 15% more than the first value, the participant is not eligible).
6. Participants should not have received bevacizumab with first-line chemotherapy or be planned to receive bevacizumab maintenance therapy.
7. Participants must be randomised within a maximum of 12 weeks from the last day of chemotherapy infusion (but no earlier than 3 weeks).

8. ECOG performance status of 0 or 1 with no deterioration over the previous 2 weeks prior to randomisation.

9, Provision, at pre-screening, of a formalin-fixed, paraffin-embedded (FFPE) tumour sample to assess tBRCA status and for HRD testing centrally. The centrally performed tBRCA test results must be available prior to randomisation and must indicate that the participant has a BRCAwt tumour, defined by the absence of a deleterious or suspected deleterious BRCA mutation by central testing.

10, Adequate organ and marrow function.

Key Exclusion Criteria:

* 1, Participants with stable disease or progressive disease on the post-treatment scan or clinical evidence of progression at the end of the participant's first-line chemotherapy treatment, or any evidence of progressive disease prior to randomization.

  2, Participant has mucinous or clear cell subtypes of epithelial ovarian cancer, carcinosarcoma, undifferentiated ovarian cancer, non-epithelial ovarian cancer, borderline tumours or low grade epithelial ovarian tumours (applies to fallopian tube and primary peritoneal tumours where applicable).

  3, Participants with Stage III disease who have had complete cytoreduction (ie, no macroscopic residual disease) at their primary debulking surgery.

  4, Participants who have undergone ˃ 2 debulking (cytoreductive) surgeries.

  5, History of another primary malignancy except for: malignancy treated with curative intent with no known active disease ≥ 5 years before the first dose of study intervention and of low potential risk for recurrence; Adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), and Stage 1, Grade 1 endometrial carcinoma. Participants with a history of localised triple negative breast cancer, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the participant remains free of recurrent or metastatic disease.

  6, Persistent toxicities (CTCAE Grade ≥2) caused by previous anticancer therapy, excluding alopecia and CTCAE Grade 2 peripheral neuropathy. Participants with irreversible toxicity that is not reasonably expected to be exacerbated by study intervention may be included after consultation with the AstraZeneca study physician.

  7, Participant is immunocompromised

  8, Prior exposure to a PARP inhibitor, including olaparib

  9, Any concurrent anticancer treatment

  10, Currently pregnant or breast-feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2026-07-27 (Estimated); Study Completion 2027-07-27 (Estimated)

PRIMARY OUTCOMES:
Superiority of olaparib as maintenance treatment relative to placebo by assessment of PFS in participants with Stage III/IV ovarian cancer with a BRCAwt HRD positive tumour and a CR/PR following standard 1st line platinum based chemotherapy treatment. | Approximately 3 years
  PFS is defined as time from randomisation until progression per RECIST 1.1 as assessed by the investigator at the local site, or death due to any cause.
Superiority of olaparib as maintenance treatment relative to placebo by assessment of PFS in participants with Stage III/IV ovarian cancer with a BRCAwt tumour and a CR/PR following standard 1st line platinum-based chemotherapy treatment. | Approximately 3 years
  PFS is defined as time from randomisation until progression per RECIST 1.1 as assessed by the investigator at the local site, or death due to any cause.

SECONDARY OUTCOMES:
Superiority of olaparib as maintenance treatment relative to placebo by assessment of OS in participants with Stage III/IV ovarian cancer with a BRCAwt HRD positive tumour and a CR/PR following standard first line platinum based chemotherapy treatment. | Approximately 4 years
  OS is defined as time from randomisation until the date of death due to any cause.
Superiority of olaparib as maintenance treatment relative to placebo by assessment of OS in participants with Stage III/IV ovarian cancer with a BRCAwt tumour and a CR/PR following standard first-line platinum-based chemotherapy treatment. | Approximately 4 years
  OS is defined as time from randomisation until the date of death due to any cause.
Superiority of olaparib as maintenance treatment relative to placebo by assessment of TFST in participants with a BRCAwt HRD positive tumour and a CR or PR following standard first-line platinum-based chemotherapy treatment. | Approximately 4 years
  TFST is defined as time from randomisation until the start date of the first subsequent anti-cancer therapy after discontinuation of randomised treatment, or death due to any cause.
Superiority of olaparib as maintenance treatment relative to placebo by assessment of TFST in participants with a BRCAwt tumour and a CR or PR following standard first line platinum based chemotherapy treatment. | Approximately 4 years
  TFST is defined as time from randomisation until the start date of the first subsequent anti-cancer therapy after discontinuation of randomised treatment, or death due to any cause.
Superiority of olaparib as maintenance treatment relative to placebo by assessment of PFS2 in participants with a BRCAwt HRD positive tumour and a CR or PR following standard first-line platinum based chemotherapy treatment. | Approximately 4 years
  PFS2 is defined as the time from the randomisation to the earliest of the progression event (following the initial progression), subsequent to first subsequent therapy or death.
Superiority of olaparib as maintenance treatment relative to placebo by assessment of PFS2 in participants with a BRCAwt tumour and a CR or PR following standard first-line platinum based chemotherapy treatment. | Approximately 4 years
  PFS2 is defined as the time from the randomisation to the earliest of the progression event (following the initial progression), subsequent to first subsequent therapy or death.
Superiority of olaparib as maintenance treatment relative to placebo by assessment of TSST in participants with a BRCAwt HRD positive tumour and a CR or PR following standard first-line platinum based chemotherapy treatment. | Approximately 4 years
  TSST is defined as time from randomisation until the start date of the second subsequent anti-cancer therapy after discontinuation of first subsequent treatment, or death due to any cause.
Superiority of olaparib as maintenance treatment relative to placebo by assessment of TSST in participants with a BRCAwt tumour and a CR or PR following standard first-line platinum based chemotherapy treatment. | Approximately 4 years
  TSST is defined as time from randomisation until the start date of the second subsequent anti-cancer therapy after discontinuation of first subsequent treatment, or death due to any cause.
Superiority of olaparib as maintenance treatment relative to placebo by assessment of time to TDT in participants with a BRCAwt HRD positive tumour and a CR/PR following standard first-line platinum based chemotherapy treatment. | Approximately 3 years
  TDT is defined as time from randomisation until discontinuation of treatment for any reason, including disease progression, toxicity and death.
To demonstrate superiority of olaparib as maintenance treatment relative to placebo by assessment of time to TDT in participants with a BRCAwt tumour and a CR or PR following standard first-line platinum based chemotherapy treatment. | Approximately 3 years
  TDT is defined as time from randomisation until discontinuation of treatment for any reason, including disease progression, toxicity and death.
Superiority of olaparib as maintenance treatment relative to placebo by assessment of time to earliest progression by RECIST 1.1/CA 125/death in participants with a BRCAwt HRD positive tumour and a CR/PR following 1st line platinum based chemotherapy | Approximately 3 years
  Time to earliest progression by RECIST 1.1/CA 125 or death will be measured from time of randomisation to the earlier date of RECIST 1.1/CA-125 progression or death by any cause.
Superiority of olaparib as maintenance treatment relative to placebo by assessment of time to earliest progression by RECIST 1.1/CA 125/death in participants with a BRCAwt tumour and a CR/PR following first-line platinum based chemotherapy. | Approximately 3 years
  Time to earliest progression by RECIST 1.1 or CA 125 or death will be measured from time of randomisation to the earlier date of RECIST 1.1 or CA-125 progression or death by any cause.
Assess Health-related quality of life in participants treated with olaparib compared with placebo in participants with a BRCAwt HRD positive tumour and a CR or PR following standard first-line platinum based chemotherapy treatment | Approximately 3 years
  Change from baseline in EORTC QLQ C30.
Assess Health-related quality of life in participants treated with olaparib compared with placebo in participants with BRCAwt tumour and a CR or PR following standard first-line platinum based chemotherapy treatment | Approximately 3 years
  Change from baseline in EORTC QLQ C30.

OTHER OUTCOMES:
Assess the safety and tolerability of olaparib in terms of AEs/SAEs as compared with placebo in participants with a BRCAwt tumour and a CR or PR following standard first-line platinum-based chemotherapy treatment. | Approximately 3 years
  Graded according to the National Cancer Institute (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, Principal Investigator — Fudan University
Locations (67):
- Chile (3):
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (30):
  - Research Site, Baoji
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jiaxing
  - Research Site, Jining
  - Research Site, Lanzhou
  - Research Site, Linyi
  - Research Site, Nanjing
  - Research Site, Qingdao
  - Research Site, Rui’an
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xuzhou
  - Research Site, Yanji
  - Research Site, Zibo
  - Research Site, Zunyi
- Colombia (2):
  - Research Site, Bogotá
  - Research Site, Medellín
- India (7):
  - Research Site, Gūrgaon
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Madurai
  - Research Site, Namakkal
  - Research Site, Nashik
  - Research Site, New Delhi
- Peru (3):
  - Research Site, Arequipa
  - Research Site, Lima
  - Research Site, San Isidro
- Russia (6):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
  - Research Site, Yekaterinburg
- Research Site, Port Elizabeth, South Africa
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Karşıyaka
  - Research Site, Samsun
- Ukraine (7):
  - Research Site, Chernihiv
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kryvyi Rih
  - Research Site, Kyiv
  - Research Site, Zaporizhzhia
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home